CLINICAL TRIAL: NCT06164314
Title: Effect of Perioperative Dexmedetomidine on Postoperative Delirium in Patients With Brain Tumors: a Randomized Placebo-controlled Trial
Brief Title: Perioperative Dexmedetomidine on Postoperative Delirium in Patients With Brain Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023064
Record Dates: First submitted 2023-11-12; First posted 2023-12-11 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dex group (Experimental): Subjects assigned to Dex group will receive a continuous dexmedetomidine infusion (0.4 ug/kg/h) after anesthesia induction until dural closure, and then received an intravenous analgesia pump with dexmedetomidine(0.08ug/kg/h), sufentanil and antiemetic until 48 hours postoperatively
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Subjects in the Placebo group were given comparable volumes of normal saline during the surgery, and intravenous analgesia pump also contains sufentanil and antiemetic, but no dexmedetomidine used until 48 hours postoperatively.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — In Dex group, dexmedetomidine will continue to be used during and after surgery, with a infusion of 0.4ug/kg/ h from anesthesia induction to dural closure, and then 0.08ug/kg/ h to 48 hours postoperatively.In placebo group, equivalent normal saline will be injected during operation, and the intravenous analgesia pump will not contain dexmedetomidine after operation

SUMMARY:
Neurosurgery is a risk factor for delirium. Dexmedetomidine might reduce delirium by reducing neuroinflammation, improving postoperative analgesia and sleep quality. The the primary hypothesis is that perioperative administration of dexmedetomidine can reduce the incidence of postoperative delirium

DETAILED DESCRIPTION:
The investigators will be required to attend the professional training before recruitment and strictly adhere to the study protocol. All the raw data will be recorded in the case report forms. Data will be entered doubly performed by two investigators and monitored securely in an electronic database with password protection at the medical center. The data base will be locked after all data have been cleaned. All the original fles will be maintained in storage for 5 years after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with temporal glioma scheduled for a elective craniotomy
* Age ≥18 years
* Obtain written informed consent.

Exclusion Criteria:

* Patients with severe preoperative cognitive impairment
* History of traumatic brain injury or previous neurosurgery
* History of psychotropic medications
* Allergy to dexmedetomidine
* Pregnant or lactating women
* History of obstructive sleep apnoea syndrome
* Severe bradycardia(heart rate <40 beats/min), sick sinus syndrome or second-to-third degree atrioventricular block
* Severe hepatic dysfunction
* Severe renal dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of delirium postoperatively | the postoperative 5 days
  Using the Confusion Assessment Method for Intensive Care Unit (CAM-ICU) for critical care patients, or the 3-min Diagnostic interview for Confusion Assessment Method (3D-CAM) for ward assessment,combined with the Richmond Agitation Sedation Scale (RASS). Delirium assessments will be only conducted in patients with RASS sedation score exceeding -4.The CAM-ICU and the 3D-CAM describes four main characteristics of delirium: acute altered mental state ,fluctuating level of consciousness, inattention, and confusion of thought. If both the first and second features are present, and both the third or fourth features are present, the patient is diagnosed with postoperative delirium.

SECONDARY OUTCOMES:
the severity of postoperative delirium | the postoperative 5 days
  Using the Delirium Rating Scale-Revised -98 (DRS-R-98) to assess.There are 3 diagnostic items (0~2 or 0~3 points each) and 13 severity assessment items (0~3 points each), for a total of 46 points. The higher the score, the more severe the delirium.
the intensity of pain | the postoperative 5 days
  Using numerical rating scale (NRS) for pain to assess, ranging from 0 to 10 points, with 10 representing the worst imaginable pain.
the quality of sleep | the postoperative 5 days
  The Richards-Campbell Sleep Questionnaire (RCSQ) will be used to assess subjective sleep quality. The scale is composed of 5 items, including sleep depth, sleep latency, wake times, return to sleep and overall sleep quality, all of which are scored by 0 ~ 100mm visual simulation (1 mm=1 point). The total score of the scale is the average score of the 5 items, and the higher the score, the better the sleep quality.
safety outcomes | from the start of medicine infusion to 48 hours postoperatively
  Safety outcomes includes the incidence of hypotension (systolic blood pressure below 95mmHg or below 30% of baseline), hypertension (systolic blood pressure above 180mmHg or 30% above baseline), bradycardia (heart rate less than 40 beats per minute), tachycardia (heart rate more than 100 beats per minute), delayed extubation (more than from the end of surgery to 2 hours after surgery, for the ICU patients (more than 4 hours),hypoxemia (SpO2<90%)

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeng M, Zheng M, Wang J, Li S, Ji N, Peng Y. Effect of perioperative dexmedetomidine on postoperative delirium in patients with brain tumours: a protocol of a randomised controlled trial. BMJ Open. 2024 Nov 7;14(11):e084380. doi: 10.1136/bmjopen-2024-084380. PMID 39515867